CLINICAL TRIAL: NCT04726072
Title: Yoga and Brain Aging
Brief Title: Kundalini Yoga & Healthy Neurological Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Davis Institute (Other)
Collaborators: Kripalu Institute and the Mind and Life Institute (Unknown)
Responsible Party: Principal Investigator, Soham Rej MD, MSc, MD, MSc, Lady Davis Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IUSMD-16-55
Record Dates: First submitted 2020-12-02; First posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Neurological Aging

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two groups for the duration of the study. One group was a Kundalini Yoga intervention while the other was a psychoeducation control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kundalini Yoga (Experimental): The Kundalini yoga intervention is a mixture of basic yoga, breathing exercises and meditation. Participants were also asked to do at-home practice for half an hour daily.
  Interventions: Behavioral: Kundalini Yoga
- Psychoeducation (Active Comparator): The psychoeducation group consisted of teaching participants about healthy aging. Participants were asked to do at-home practice for half an hour daily
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Kundalini Yoga — Participants met once a week for two hours for 12 weeks total. The Kundalini yoga intervention is a mixture of basic yoga, breathing exercises, and meditation. Participants were also asked to do at-home practice for half an hour daily.
  Arms: Kundalini Yoga
Behavioral: Psychoeducation — Participants met once a week for two hours for 10 weeks total. The psychoeducation group acted as our control group and consisted of teaching participants about healthy aging. Participants were asked to do at-home practice for half an hour daily.
  Arms: Psychoeducation

SUMMARY:
This randomized-control trial pilot study investigates the potential neuroprotective effects of mindfulness-based interventions in older adults. In this study, the researchers examine the effects of Kundalini yoga on neurotypical brain aging with a focus on volumetric changes in the bilateral hippocampi and posterior cingulate cortex. 14 healthy, meditation-naïve participants (ages 60 to 80) were recruited. Half were randomly assigned to the Kundalini yoga group and half to the psychoeducation group. Overall, three participants withdrew from the study. The yoga intervention lasted for 12 weeks and the psychoeducation intervention lasted for 10 weeks. Structural and functional Magnetic Resonance Imaging (MRI) data were obtained at baseline and 12-week follow-up. The researchers will focus on analyzing structural MRI data, examining gray matter volume within a priori regions of interest (bilateral hippocampi and posterior cingulate cortex). Results from this pilot study are intended to provide effect-size estimates for future studies that would confirm the effects of Kundalini yoga on neurological aging. Researchers predict participation in the Kundalini yoga intervention, compared to the psychoeducation control condition, will result in a greater increase in gray matter volume of the bilateral hippocampi and posterior cingulate cortex from pre- to post-intervention. If the results are positive, this would provide initial neurobiological support for Kundalini yoga as a potential means to mitigate the effects of neurological aging and as a preventive measure for Alzheimer's disease and dementia, which could be assessed in future confirmatory clinical trials.

DETAILED DESCRIPTION:
Recruitment:

Participants were recruited from the Douglas Hospital as well as from the broader community through the use of an advertisement in The Gazzette and Le Devoir newspapers. Participants were pre-screened to ensure they were eligible for the study based on the inclusion and exclusion criteria. This screening process included a cognitive assessment as well as having participants lie in a mock scanner to assess their level of comfort and ability to complete the neuroimaging scans required for the study. If anyone was unable to comfortably lie in the mock scanner, then they were still given the option to participate in the program, but not as a research participant. A total of 14 participants were recruited for the study.

Intervention Groups:

Participants were evenly and randomly assigned to one of two groups. One group was the Kundalini yoga group while the other was a psychoeducation program (which acted as the control group). All seven participants in the Kundalini yoga group completed the study while only four participants in the psychoeducation group completed the study (i.e. three participants withdrew from the study). Participants were between the ages of 60 to 80 years old with no prior meditation experience and were relatively healthy with a baseline Mini-Mental State Examination score of 28-30. Participants were matched across groups for gender, age, and years of education. The study lasted about 12 weeks for participants in the Kundalini yoga group and about 10 weeks for those in the control group. The discrepancy in program length was the result of scheduling complications. Each condition had weekly, two-hour, group-based sessions that were led by a trained interventionist. The Kundalini yoga group exercises were customized for participants to ensure safety and are a mixture of postures, breathing exercises, and meditation. Additionally, participants were encouraged to do practice exercises at-home for half an hour a day. They were asked to report on the extent of their at-home practices. The control group consisted of a psychoeducation program where participants were taught about memory and healthy aging. Participants in this group were also encouraged to do at home tasks for about half an hour a day.

Data Collection:

Structural and functional MRI data were obtained both before and after participating in the intervention. The order of scanning was randomized and counterbalanced within and across subjects. Overall, scanning lasted about one hour in duration.

During the structural scan, participants were asked to lie down for 10 minutes. There were no images presented on the screen during this time. For the resting-state functional scan, participants were asked to look at a fixation cross presented on the screen while trying to relax.

Acquisition Parameters of both Structural and Functional Scanning:

Structural

* Orientation: Coronal
* Phase enc. dir.: R>>L
* # of slices: 320
* FoV: 206 mm IS x 320 RL
* Slice thickness:$$0.64mm isotropic
* TR: 2500ms
* TE: 198ms
* PAT mode: GRAPPA
* Accel. factor: 2
* Ref. lines PE: 24
* Band width: 710 Hz/Px
* Echo spacing: 4ms
* Scan time: 10:02 minutes
* Coil elements:$$HEA;HEP

Resting-State

* # of slices: 32
* Orientation: Transversal ACBPC
* Phase enc. dir.:A>>P
* FoV: 128 mm IS x 256 mm AP
* Motion correction = off
* Slice thickness: 4mm
* TR: 2000ms
* TE: 30ms
* Flip angle: 90°
* PAT mode: none
* Band width: 2442 Hz/Px
* Echo spacing: 0.47ms
* GLM statistics = off
* # of measurements: 150
* Scan time: 5:04 minutes
* Coil elements: HEA;HEP

ELIGIBILITY:
Inclusion Criteria:

* Neurologically Healthy
* Between ages 60-80 years old
* Little to no meditation experience

Exclusion Criteria:

* Any neurological or psychiatric disorder or a family history of such disorders
* Uncomfortable or unable to undergo MRI scanning
* Diabetes, or a cardiovascular or respiratory illness
* Regular alcohol or tobacco consumption

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2018-04-24 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Gray Matter Volume in Bilateral Hippocampi and Posterior Cingulate Cortex at 10-12 weeks | Structural neuroimaging scans were taken at baseline (0 weeks) and post-intervention (10 to 12 weeks, 10 weeks for the control group and 12 weeks for the Kundalini Yoga intervention group).
  Participants were placed in an MRI machine to conduct structural imaging scans to determine the potential impact of the intervention on gray matter volume in bilateral hippocampi and posterior cingulate cortex of participants after the intervention (10-12 weeks from baseline; 10 weeks for the psychoeducation control group and 12 weeks for the Kundalini yoga intervention. Discrepancy in intervention durations was a result of scheduling conflicts).Voxel-Based Morphometry was used to analyze structural images.

SECONDARY OUTCOMES:
Change from Baseline Functional Connectivity in the Posterior Cingulate Cortex at 10-12-weeks. | Functional neuroimaging scans were taken at baseline (0 weeks) and post-intervention (10-12 weeks; 10 weeks for the psychoeducation control group and 12 weeks for the Kundalini yoga intervention).
  Participants were placed in an fMRI machine to conduct resting-state functional imaging scans (each resting state acquisition lasted 5:04 minutes) to determine the potential impact of the intervention on functional connectivity in the posterior cingulate cortex of participants after the intervention (10-12 weeks from baseline; 10 weeks for the psychoeducation control group and 12 weeks for the Kundalini yoga intervention. Discrepancy in intervention durations was a result of scheduling conflicts).

CONTACTS AND LOCATIONS:
Overall Officials: Soham Rej, MD, MSc, Principal Investigator — Lady Davis Research Institue
Locations (1):
- Douglas Mental Health University Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No